CLINICAL TRIAL: NCT05557721
Title: Uddevalla Skövde Transscleral Micropulse Study: Efficacy and Safety of Micro Pulse Transscleral Laser Treatment (MP-TLT) in Glaucoma Patients Performed in Topical Lidocaine Anaesthesia
Brief Title: Uddevalla Skövde Transscleral Micropulse Study
Acronym: USTMS
Status: Enrolling by invitation | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: USTMS; 278487 (Registry Identifier: FoU i VGR)
Record Dates: First submitted 2022-09-19; First posted 2022-09-28 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Primary Open Angle Glaucoma; Pseudoexfoliation Glaucoma
Keywords: Micro pulse transscleral laser treatment (MP-TLT)
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome | interventions — Lidocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MP-TLT in topical anesthesia: Patients will receive topical anesthesia with tetracaine hydrochloride 1% three times, 5 minutes apart. Then, lidocaine gel 2% will be applied on the surface of the eye and refilled as needed for 10 minutes, as well as manipulated for a good coverage. Thereafter, MP-TLT will be performed with the Iridex CycloG6 laser with the revised P3 probe, according to the recent consensus recommendations. In brief, this includes MP-TLT with 2500 mW, 31.3% duty cycle, four 20 second sweeps per hemisphere, avoiding the 3 and 9 o'clock meridians and sectors with scleral thinning.
  Interventions: Procedure: Topical lidocaine; Procedure: MP-TLT

INTERVENTIONS:
Procedure: Topical lidocaine — Patients will receive topical anesthesia with tetracaine hydrochloride 1% three times, 5 minutes apart. Then, lidocaine gel 2% will be applied on the surface of the eye and refilled as needed for 10 minutes, as well as manipulated for a good coverage.
Procedure: MP-TLT — Micro pulse transscleral laser treatment will be performed with the Iridex CycloG6 laser with the revised P3 probe, according to the recent consensus recommendations.
  In brief, this includes MP-TLT with 2500 mW, 31.3% duty cycle, four 20 second sweeps per hemisphere, avoiding the 3 and 9 o'clock meridians and sectors with scleral thinning.

SUMMARY:
Micro pulse transscleral laser treatment (MP-TLT) is a relatively new method to reduce the intraocular pressure (IOP) in glaucoma. New recommendations regarding the treatment protocol has recently been developed and was published 2022.

The overall objective is to evaluate the efficacy and safety of the proposed treatment method in an independent study. In addition, the outcome of MP-TLT in patients with pseudoexfoliation glaucoma, which is relatively common in the Nordic countries, and primary open angle glaucoma will be studied separately.

The IOP change over the course of one year will be monitored, as well as success rate and survival. Further, patient-reported discomfort from the treatment and the occurrence of any adverse events or complications will be studied.

DETAILED DESCRIPTION:
Forty patients scheduled for MP-TLT by their ophthalmologist will be recruited. One eye per patient is included, based on randomization, even if both are treated. MP-TLT will be performed according to the current recommendations.

Baseline IOP will be calculated as the mean of three separate measurements taken on different days preoperatively. IOP will then be measured 1 week, 1 month, 3 months, 6 months and 12 months after MP-TLT.

The central corneal thickness (CCT), the central retinal thickness (CRT), anterior chamber flare and the visual field (HFA 24-2 faster) will also be measured preoperatively and during follow up.

In accordance with the World Glaucoma Association guidelines, no adjustment for multiple comparisons is planned in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open angle glaucoma (POAG) or pseudo exfoliative glaucoma (PXFG)
* Age ≥ 18 years
* The patient is expected to be able to adequately undergo and cooperate in the treatment and follow-up as described in the study protocol.
* The patient is judged to have good compliance with already prescribed pharmacological glaucoma treatment.

Exclusion Criteria:

* Allergy or hypersensitivity to tetracaine or lidocaine
* Prior transscleral laser or cryo treatment.
* Prior eye surgery (including intravitreal injection) or pressure-lowering laser treatment (SLT/ALT/MDLT) during the last 2 months.
* Planned or expected eye surgery (eg., cataract surgery or intravitreal injection) in the coming year.
* History of macular edema.
* History of corneal edema.
* History of uveitis during the past year.
* Existing thinning in the sclera of a greater extent than 30 degrees (one "clock-hour") of the circumference.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients referred for MP-TLT at the ophthalmology departments of the NU Hospital Group and the Skaraborg Hospital are recruited sequentially.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Relative IOP change (percent) | 6 months
  Relative IOP (intraocular pressure) change (percentage relative to baseline) for the entire study population. "Last observation carried forward" will be used in cases with treatment escalation or reduction during follow up. Patients with peroral glaucoma treatment at baseline are not included in this analysis.
Relative IOP change (percent) for POAG and PXFG eyes separately | 6 months
  Relative IOP change (percentage relative to baseline) for the eyes with a diagnosis of primary open angle glaucoma, or pseudo exfoliative glaucoma, respectively. "Last observation carried forward" will be used in cases with treatment escalation or reduction during follow up. Patients with peroral glaucoma treatment at baseline are not included in this analysis.
Perioperative pain on a visual analogue scale (VAS) | Immediately after surgery
  The patient will report pain during MP-TLT treatment on a VAS immediately after surgery.
  A 10 cm horizontal line without markings will be presented. One end of the line represents "no pain" and the other "worst imaginable pain". The patient marks the position on the scale that corresponds to the level of perceived pain. The number of millimeters from the "no pain" end is the result. Higher is worse.
  If there was a need for supplementary anesthesia, the grading applies to the experience before supplementation.

SECONDARY OUTCOMES:
Success proportion after 12 months | 12 months
  Eyes will be graded with either "success" or "failure" after one year of follow up. Definition of success (all must be fulfilled):
  * Reduction of the IOP by at least 20% compared to baseline and/or reduction in pharmacological glaucoma treatment.
  * IOP ≥ 6 mmHg
  * No additional IOP reducing intervention performed after MP-TLT.
Survival | 12 months
  Kaplan-Meier survival analysis regarding achievement and maintenance of "success" as defined above.
Relative change (percent) of the IOP 1 week, 1 month, 3 months and 12 months after MP-TLT. | 12 months
  IOP change relative to baseline 1 week, 1 month, 3 month and 12 months after MP-TLT. "Last observation carried forward" will be used in cases with treatment escalation or reduction during follow up. Patients with peroral glaucoma treatment at baseline are not included in this analysis.
Postoperative pain on a VAS 1 hour, 5 hours, and 24 hours postoperatively | 1 hour, 5 hours, and 24 hours postoperatively
  Postoperative pain on a VAS 1 hour, 5 hours, and 24 hours postoperatively. See above for further description.
Patient reported discomfort on an arbitrary scale | 1 month
  The patients will report peri- and postoperative pain, postoperative light sensitivity, visual impairment and hyperemia. The scale goes between 0 (no sensation) and 4 (worst imaginable). The scale was developed for the OSLT trial (NCT03798223). Comparisons will be made with the results from that trial.
Change in central retinal thickness (CRT) postoperatively | 3 months
  The thickness in the central retinal field will be measured with optical coherence tomography (OCT) at baseline and 1 week, 1 month and 3 months postoperatively. The relative change (percent) will be calculated for each time point.
Change in central corneal thickness (CCT) postoperatively | 1 month
  The central corneal thickness (CCT) in the thinnest point will be measured with Pentacam at baseline and 1 week and 1 month postoperatively. The relative change (percent) will be calculated for each time point. Applies only to NU patients (one of the centers).
Change of flare in the anterior chamber postoperatively | 1 month
  Flare in the anterior chamber will be measured with a Kowa laser flare meter at baseline and 1 week and 1 month postoperatively. The relative change (percent) will be calculated for each time point. Applies only to SkaS patients (one of the centers).
Change in visual field index (VFI) during follow-up | 12 months
  The visual field will be assessed with a Humphrey field analyzer (HFA) 24-2 faster at baseline and then 1 and 12 months postoperatively. The change in VFI, expressed in percentage points, will be calculated for each time point.
Adverse events | 12 months
  Suspected adverse events will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Dahlgren, MD, Principal Investigator — Vastra Gotaland Region; Marcelo Ayala, MD, PhD, Study Chair — Vastra Gotaland Region
Locations (2):
- Sweden (2):
  - Department of Ophthalmology, Skaraborg Hospital, Skövde, Västra Götaland County
  - Department of Ophthalmology, NU Hospital Group, Uddevalla, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grippo TM, de Crom RMPC, Giovingo M, Toteberg-Harms M, Francis BA, Jerkins B, Brubaker JW, Radcliffe N, An J, Noecker R. Evidence-Based Consensus Guidelines Series for MicroPulse Transscleral Laser Therapy: Dosimetry and Patient Selection. Clin Ophthalmol. 2022 Jun 7;16:1837-1846. doi: 10.2147/OPTH.S365647. eCollection 2022. PMID 35698599